CLINICAL TRIAL: NCT05477654
Title: TwinBrain Parkinson's Disease Clinical Trial
Brief Title: Motor-cognitive Dual-task in Healthy Older Adults and Early Parkinson's Disease Patients
Acronym: TwinBrainPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Science and Research Centre Koper (Other)
Collaborators: Technische Universität Berlin (Other); University of Geneva, Switzerland (Other); University of Trieste (Other); University Maribor (Other)
Responsible Party: Principal Investigator, Marusic, Associate professor, Science and Research Centre Koper
Other Study IDs: TwinBrainPDstudy
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Parkinson Disease; Motor Disorders; Cognitive Impairment
MeSH Terms: conditions — Parkinson Disease; Motor Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's disease patients: Patients with an early diagnosis of Parkinson's disease
  Interventions: Diagnostic Test: Extensive motor-cognitive testing protocol
- Healthy controls: Healthy controls who are age-matched
  Interventions: Diagnostic Test: Extensive motor-cognitive testing protocol

INTERVENTIONS:
Diagnostic Test: Extensive motor-cognitive testing protocol — Screening of their functional performance while monitoring brain and muscle activity

SUMMARY:
Neuromuscular dysfunction is common in older adults and even more pronounced in neurodegenerative diseases. In Parkinson's disease (PD), a complex set of factors often prevents effective performance of activities of daily living that require intact and simultaneous performance of motor and cognitive tasks. In the current study we aim at employing the Mobile Brain/Body Imaging approach (MoBI) to gain further insides of neuromuscular biomarkers revealing the decrements of older adults with an early PD. The cross-sectional study will be evaluated through the multifactorial mixed-measure design.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for the healthy older participants will be:

* no diagnosis of cognitive or movement disorder,
* score > 7 for the Short Physical Performance Battery (SPPB),
* living independently in the community,
* age range between 55 and 70 years,
* no color blindness.

Inclusion criteria for the early-stage PD patients:

* diagnosed according to the last MDS criteria (2015),
* duration of the disease less than 5 years,
* positive DATSCAN,
* diagnosed akinetic-rigid or mixed phenotype,
* score of 1 or maximally 2 on the Hoehn and Yahr scale (Hoehn & Yahr, 1967),
* MoCA score ≥ 24 points,
* score > 7 for the SPPB,
* age range between 50 and 75 years,
* no color blindness
* living independently in the community.

Exclusion Criteria:

* advanced stages of PD (Hoehn and Yahr score > 2)
* any acute or chronic diseases, especially of the peripheral and central nervous system, heart failure, respiratory failure, severe osteoarthritis, and major psychiatric illness such as depression
* MoCA score < 24 points,
* severe disabling tremor,
* recurrent falls,
* impaired vision that is not corrected with e.g., glasses,
* low SPPB score

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include healthy age-matched controls and patients with an early diagnosis of Parkinson's disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
dual-task costs while walking | Day 1
  Test for dual-task costs associated with the concurrent execution of overground walking and a secondary cognitive task
dual-task costs while standing | Day 1
  Test for dual-task costs associated with the concurrent execution of semi-tandem stance and a secondary cognitive task
dual-task costs while execution of isometric task | Day 1
  Test for dual-task costs associated with the concurrent execution of isometric contraction and a secondary cognitive task

SECONDARY OUTCOMES:
The Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Day 1
  Assessment of various aspects of PD including motor and non-motor experience of daily living and the related complications

CONTACTS AND LOCATIONS:
Locations (1):
- Science and research centre Koper, Koper, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marusic U, Peskar M, Somen MM, Kalc M, Holobar A, Gramann K, Wollesen B, Wunderlich A, Michel C, Miladinovic A, Catalan M, Buoite Stella A, Ajcevic M, Manganotti P. Neuromuscular assessment of force development, postural, and gait performance under cognitive-motor dual-tasking in healthy older adults and people with early Parkinson's disease: Study protocol for a cross-sectional Mobile Brain/Body Imaging (MoBI) study. Open Res Eur. 2023 Nov 10;3:58. doi: 10.12688/openreseurope.15781.3. eCollection 2023. PMID 38009088